CLINICAL TRIAL: NCT05175092
Title: Neo-adjuvant Chemotherapy Plus Living Donor Liver Transplantation (LDLT) for Non-Resectable Liver Metastases From Colorectal Cancer (CRC)
Brief Title: Living Donor Liver Transplantation for CRC Liver Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0021; 2021-0021 (Other: HSIRB UW Madison); A539742 (Other: UW Madison); Protocol Version 7/15/2022 (Other: UW Madison); UW20113 (Other: UWCCC OnCore ID)
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2023-11

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: living donor liver transplant

STUDY DESIGN:
Intervention Model Description: single-center, open-label, two-stage recruitment
  * pilot study of 5 recipients to determine if LDLT is a suitable treatment for patients with non-resectable LM with 3 years of follow-up, if Overall Survival greater than 60%, then
  * stage two recruitment focusing on accruing additional recipients will commence.
  * control group of participants that sign the informed consent and are enrolled in the study but do not undergo LDLT due to a lack of an eligible donor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intent to Treat: LDLT (Experimental): Living Donor Liver Transplantation
  Interventions: Procedure: Living Donor Liver Transplantation
- Control Group (No Intervention): Enrolled but does not receive LDLT

INTERVENTIONS:
Procedure: Living Donor Liver Transplantation — The LDLT will be performed by the UW Division of Transplantation in accordance with the standard of care for this operation.
  Other Names: LDLT
  Arms: Intent to Treat: LDLT

SUMMARY:
This study will test the safety and efficacy of living donor liver transplant after standard-of-care chemotherapy for participants with non-resectable liver metastases (LM) from colorectal cancer. 25 donor-recipient pairs will be enrolled (50 participants). Donors will be on study for 2 years and recipients will be on study for up to 5 years.

DETAILED DESCRIPTION:
This study is a single center, open-label study available to male and female adults with CRC LM that are deemed to be "unresectable" and who are receiving standard of care chemotherapy. Participants will be worked up for LDLT while continuing to receive chemotherapy and, if deemed eligible for surgery, will stop chemotherapy 4 weeks prior to receiving a living donor transplant. Recipients will be followed for 5 years (for safety, survival and disease recurrence for purposes of study data collection). They will continue to be monitored for safety, survival and disease recurrence indefinitely as part of University of Wisconsin (UW) Health's Organ Transplant Program care standards. Living liver donors will be followed for 2 years after transplant surgery for safety monitoring as part of this study.

Recruitment will be done in two stages. The first stage will be a pilot study of 5 recipients to determine if LDLT is a suitable treatment for patients with non-resectable LM. If, after 3 years of follow-up, the overall survival is greater than 60%, stage two recruitment will commence. Thus, an interim analysis will be done for the first 5 recipients prior to requiring a larger number of subjects. Stage two recruitment will focus on accruing a total of up to 20 additional recipients to be analyzed.

The control group will consist of any potential recipients that sign the informed consent and are enrolled in the study but do not undergo LDLT due to a lack of an eligible donor. These participants will be referred back to their medical oncologists to receive standard of care chemotherapy, and will continue to be followed as the control group.

Patients who sign the informed consent and are enrolled in the study with an eligible live donor but do not undergo LDLT due to disease progression or a contraindication is established for undergoing LT (exclusion criteria) will also be referred back to their medical oncologists to receive standard of care chemotherapy. This group will be followed as part of the intent to treat cohort.

ELIGIBILITY:
Recipient Inclusion Criteria

In order to be eligible to participate in this study, a potential recipient must meet all of the following criteria prior to transplant procedure:

* General inclusion criteria:

  * Male or female, aged 18 - 65 years old inclusive, at study entry
  * Willing and able to provide written informed consent
  * Reside in the United States
  * Negative serum pregnancy test for women of childbearing potential
* Cancer-related inclusion criteria:

  * Eastern Cooperative Oncology Group (ECOG) : 0 or 1 at all times prior to LDLT
  * Biopsy-proven colorectal LM
  * Tumor must have the following characteristics

    * Non-resectable LM (by consensus of three hepatobiliary (HPB) surgeons). All potential recipients will be presented at Multidisciplinary Tumor Rounds for discussion of treatment options
    * Synchronous or Metachronous disease
    * R0 resection can be achieved by total hepatectomy
    * Primary CRC tumor stage is ≤T3 and ≤N2
    * Oslo score of 0-1. The Oslo Score summarizes 4 negative predictive factors for overall survival after liver transplantation for CRLM where each factor is assigned 1 point; maximal diameter of the largest lesion >5.5 cm, pre-transplant CEA level >80 μg/L, progressive disease at time of liver transplant and interval from diagnosis to transplant <2 years
    * The patient has undergone first-line "standard of care" chemotherapy for a minimum of 3 months (at the time of screening), with demonstrated stability or regression of LM based on RECIST v 1.1 criteria
    * The only site of metastases is the liver (Staging CT scans are clear of metastases)
* Transplant related inclusion criteria:

  * At least one ABO compatible living donor has been identified, and has completed an intake history which, upon review by the Living Donor team, is deemed acceptable and demonstrates no obvious contraindications to donation (Altruistic donors will not be accepted for the study).
  * Complete colonoscopy within the 12 months prior to potential recipient's inclusion, showing no signs of local recurrence
  * Prior authorization by private insurance as a single payer exception is required. This will be discussed on a case-by-case basis with the insurance providers and the Transplant Financial Group
  * Creatinine clearance greater than or equal to 50 ml/min
  * Absolute neutrophil count greater than or equal to 1,500/uL
  * Child-Pugh score of A
  * Meets criteria to undergo a liver transplantation

Recipient Exclusion Criteria:

A potential recipient who meets any of the following criteria will be excluded from participation in this study:

* General exclusion criteria:

  * Substance abuse, medical, psychological or social conditions that may interfere with the potential recipient's participation in the study or evaluation of the study results
  * Known or suspected allergy to any agent given in association with this trial
  * Any condition that is unstable or which could jeopardize the safety of the potential recipient and his/her compliance in the study
  * Pregnant or breast-feeding patients
* Cancer-related exclusion criteria:

  * Previous or concurrent cancer that is distinct in primary site or histology from adenocarcinoma, except ductal carcinoma in situ, cervical carcinoma in situ, localized prostate cancer, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated 5 years prior to entry is permitted
  * Progression of LM at any time point prior to transplant surgery
  * LM show no major vascular invasion: no vena cava involvement and no porta hepatis involvement as seen on scans (including PET-CT), or through endoscopic ultrasound and exploratory laparotomy sampling of porta hepatis lymph nodes
  * BRAF+ mutation or microsatellite instability of either primary tumor or LM
* Transplant-related exclusion criteria:

  * Renal dysfunction with an estimated creatinine clearance of less than 50 ml/min
  * Pulmonary insufficiency (history of chronic obstructive pulmonary disease and FEV1 /FVC < 75%)
  * History of cardiac disease:

    * Congestive heart failure > New York Heart Association (NYHA) class 2
    * Non-revascularized coronary artery disease
    * Uncontrolled hypertension (two systolic blood pressure readings greater than 150 in past 2 visits)
  * Uncontrolled infection(s) as defined per surgeon, subject may be on antibiotics at time of transplant
  * Severe liver dysfunction (Child-Pugh Score of B or C will be excluded)
  * History of solid organ transplantation

Donor eligibility criteria:

In order to be eligible to participate in this study, a potential donor must meet all of the following criteria prior to transplant procedure:

* Willing and able to provide informed consent
* Upon review by the Living Donor team, is deemed acceptable and demonstrates no obvious contraindications to donation
* Not an altruistic donor
* Before transplant surgery, must be approved as a liver donor by UW Health Transplant Program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | participants followed up to 5 years
  Overall survival, defined as length of time from the start of (neoadjuvant) chemotherapy that subjects diagnosed with colorectal liver metastases are still alive.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | up to 5 years
  DFS, defined as length of time after LDLT during which no disease is found according to RESIST v1.1 criteria.
Site of Recurrence (Organs Affected) | up to 5 years
  Patterns of recurrence will be investigated, assessed by standard of care chest, abdominal and pelvis imaging.
Number of Sites of Recurrence per Participant | up to 5 years
  Patterns of recurrence will be investigated, assessed by standard of care chest, abdominal and pelvis imaging.
Survival Rate | up to 5 years
  Surviving number of recipients who receive LDLT vs. control subjects will be assessed at 1-, 3-, and 5-years.
Quality of Life Survey Score: EORTC QLQ-C30 | up to 5 years
  Quality of life is measured at 1-, 3-, and 5-years using the EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). The questionnaire assesses multi-item scales, each item scoring from 1 to 4, with higher scores representing a higher level of symptomatology or problems.
Quality of Life Survey Score: EORTC QLQ-LMC21 | up to 5 years
  Quality of life is measured at 1-, 3-, and 5-years using the EORTC QLQ-LMC21 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). The questionnaire assesses multi-item scales, each item scoring from 1 to 4, with higher scores representing a higher level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: David P Al-Adra, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No